CLINICAL TRIAL: NCT06697977
Title: Effects of Phytosterol Supplementation on Serum Lipid Profile, Liver Enzymes, Insulin, Adiponectin, and Inflammatory Status in Patients with Nonalcoholic Fatty Liver Disease
Brief Title: Effects of Phytosterol Supplementation on Liver Function and Inflammatory Status in Patients with Nonalcoholic Fatty Liver Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Shatha Hammad, Assistant Professor, Assistant professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19/2022/458
Record Dates: First submitted 2024-10-29; First posted 2024-11-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: NAFLD; Insulin Resistance; Metabolic Syndrome; Obesity; Diabetes; Nash; Dyslipidemias
Keywords: phytosterols; NAFLD; Plant sterols; insulin; lipid profile
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Metabolic Syndrome; Obesity; Diabetes Mellitus; Dyslipidemias | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Dietary Supplement: phytosterols
- control group (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: phytosterols — 2 grams of phytosterols given as 7 pills per day
  Arms: treatment group
Dietary Supplement: placebo — placebo 7 pills per day
  Arms: control group

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is considered one of the most common chronic liver diseases worldwide, it recently became a worldwide problem with high morbidity which requires further attention. The use of natural bioactive products such as phytosterols have shown anti-NAFLD effect with little to no side effects when used as a supplement in the therapeutic protocol of NAFLD, in many animals, and In vitro studies.

Although the positive impacts of phytosterols on the prevention of hypercholesterolemia and improving liver functions have been reported in previous studies, further clinical experiments, especially human studies are needed to assure the effectiveness of phytosterols on improving liver enzymes, lipid profile, and insulin response in patients with NAFLD. In this study, we focus on the efficacy of phytosterol in a dose similar to the therapicutic lifestyle changes diet (TLC) recommendation with an aim to include it in the therapeutic protocol for NAFLD and to study the effect of some confounders that were excluded in previous studies on this relationship.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, parallel experimental trial will be conducted to explore the therapeutic potential of phytosterol supplementation against NAFLD. Patients with NAFLD will be recruited from Jordan University Hospital, Department of Gastroenterology and Hepatology.

Forty adult patients, males and females, aged less than 70, who are diagnosed with NAFLD by liver ultrasonography, and who are willing to participate will be invited to join the clinical trial and will be informed that they can leave the study whenever they want.

Participants with any history of liver transplantation, tested positive for any type of hepatitis, autoimmune hepatitis, alcohol consumption, current corticosteroids or antibiotics consumption, rapid weight loss, heart failure, renal disease, pregnant and lactating women, patients with BMI higher than 40, or who have unintentional weight loss of 5%, and patients who are consuming other supplements within three months of the study will be excluded.

A specialized physician will examine the patients, confirm the diagnosis, and ensure that all volunteers fit the inclusion criteria.

The 40 patients will be randomly divided into two groups, using a random number generator at randomization.com; the phytosterols group (n=20), who will receive capsulated 2.0g oral phytosterol powder which will be consumed with meals daily, and the control group (n= 20) who will receive a placebo capsule (microcrystalline cellulose) of 2.0g daily. Each intervention will extend for two months, and the actual intervention phases will be preceded by a 2-week run-in period, in which the participants will be asked to refrain from the consumption of high stanols and sterols in their diets.

For the entire duration of the study, patients will follow their habitual diets but will be advised to avoid high-fat foods, their physical activity will also be monitored and data on both dietary habits and physical activity will be assessed at baseline (week 0) and after the end of the study (week 8). All participants will be asked to come to the clinics every 2 weeks to collect their supplements and fill in the required questionnaires and supplement consumption checklist.

ELIGIBILITY:
Inclusion Criteria:

* any patient with NAFLD or NASH that has been diagnosed by any type of imaging.
* ability to swallow pills.
* ability to take the supplement for 3 months.

Exclusion Criteria:

* history of liver transplantation.
* tested positive for any type of hepatitis.
* diagnosed with autoimmune hepatitis.
* significant alcohol consumption.
* current corticosteroids or antibiotics consumption.
* rapid unintentional weight loss.
* diagnosed with heart failure.
* diagnosed with renal disease.
* pregnant and lactating women.
* patients with a BMI higher than 40.
* patients who are consuming other supplements within the last three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
lab tests | from enrollment to the end of 3 months
  liver enzymes (ALT, AST, GGT, ALK, Total protein, Direct bilirubin, Total bilirubin) mg/dl
lab tests | from enrollment to the end of 3 months
  lipid profile (Cholesterol, HDL, LDL, TG) mg/dl
lab tests | from enrollment to the end of 3 months
  insulin
lab tests | from enrollment to the end of 3 months
  CRP
lab tests | from enrollment to the end of 3 months
  adiponectin

SECONDARY OUTCOMES:
Anthropometric measures | from enrollment to the end of 3 months
  weight in kilograms
Anthropometric measures | from enrollment to the end of 3 months
  waist circumference by centimetre
Vital signs | from enrollment to the end of 3 months
  blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan, Amman, Jordan